CLINICAL TRIAL: NCT06651294
Title: Efficacy and Safety of Neorenal Forte as Adjuvant Treatment for the Complete Elimination of Residual Fragments After Flexible Ureterorenoscopy With Laser Lithotripsy for Renal Calculi.
Brief Title: Efficacy of Neorenal Forte for the Complete Elimination of Residual Fragments
Acronym: NERFA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Neopharm Bulgaria Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NERFA 2501-lit-002
Record Dates: First submitted 2024-10-18; First posted 2024-10-21 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-10

CONDITIONS: Urolithiasis
Keywords: Elimination of residual fragments; Flexible ureterorenoscopy; Renal calculi; Phytotherapeutic extracts
MeSH Terms: conditions — Urolithiasis; Kidney Calculi

STUDY DESIGN:
Intervention Model Description: Prospective, multicenter, double-blind, placebo-controlled, randomized, parallel-arm clinical study
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Investigators will be provided with coded products which are identical in appearance. Each individual involved in the study will be blinded to the treatment assignment until study completion. Considering the established safety profile of the formula of phytotherapeutic extracts, emergency unblinding of treatment assignment will not be necessary. So no copies of the treatment assignments will be stored at the enrollment sites. No information about the subjects will be shared with the company conducting the randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neorenal Forte (Experimental): Up to Day 10 after the endourological procedure - 2 tablets 2 times daily Followed by 80 days after end date of 2X2 dose - 1 tablet 2 times daily
  Interventions: Dietary Supplement: Neorenal Forte
- Placebo (Placebo Comparator): Up to Day 10 after the endourological procedure - 2 tablets 2 times daily Followed by 80 days after end date of 2X2 dose - 1 tablet 2 times daily
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Neorenal Forte — This specialized formulation of phytotherapeutic extracts consists of proprietary Betula pendula leaves dry extract, Herniaria glabra, Viburnum opulus, Elymus (Agropiren) repens. The product contains supplementary ingredients: microcrystalline cellulose, povidone, magnesium stearate, colorant film (brilliant blue FCF, iron dioxide).
  Arms: Neorenal Forte
Dietary Supplement: Placebo — The placebo product will be identical to the active form and will have the same composition but without the proprietary extract from Betula pendula, Herniaria glabra, Viburnum opulus, Elymus (Agropiren) repens.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy of a specialized formula of phytotherapeutic extracts (Neorenal Forte) aiding the complete elimination of residual fragments after fURS in adults.

DETAILED DESCRIPTION:
The study is being initiated to support the informed decision making by healthcare specialists on the initiation of a specific and safe formula of phytotherapeutic extracts with duration at least three months after endourological procedures, as a routine part of urolithiasis treatment, aiding the complete elimination of residual fragments, which will allow minimizing of the short-term and long-term complications.

By evaluating the percentage of complete elimination of residual fragments or fragments < 2 mm in diameter, we aim to estimat the efficacy and safety of Neorenal Forte.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 18 to 65 years of age.
2. The subject has signed informed consent approved by an Ethics Committee and agrees to the on-site study visits.
3. A stone confirmed by NCCT of kidney, ureter and urinary bladder for assessment of size, number, location and stone density, within 90 days of fURS.
4. Single or multiple kidney stones with total size of 10x10 mm to 15x10 mm.
5. Stone density 1001 - 1400 Hounsfield units (HU).
6. Subjects post fURS for laser lithotripsy of kidney stone.
7. Residual fragments < 4 mm after fURS confirmed by ultrasound on first postoperative day.
8. Subjects post one fURS.
9. fURS uncomplicated by perforation of ureter, mucosal exfoliation, damage to kidney or urinary bladder, serious bleeding or other complications.
10. No recent ureterorenoscopy within the last 6 months.
11. Body mass index 17.0 - 29.99 kg/m2 118
12. In Investigator's opinion, the subject can comply with the visit schedule and the treatment regimen and is capable of completing the study.
13. The subject has a smartphone and is capable of using it.

Exclusion Criteria:

1. Subjects with anatomical anomalies revealed by ultrasound - stenosis of the pyelo-ureteral junction, horseshoe kidney, kidney malrotation, calyceal diverticulum, and others.
2. Ureteral stenosis.
3. History of ipsilateral renal surgery.
4. Hydronephrosis.
5. Permanent JJ stent.
6. Any conditional or absolute contraindications for fURS.
7. Combined ipsilateral stone in the ureter or contralateral stone in the upper urinary canal or a stone in the lower urinary canal, requiring simultaneous surgery.
8. Subjects with positive urine culture, until resolution.
9. History of endourological intervention (e.g. nephrostoma, ureteral catheter) before fURS.
10. Stone density <1000 and >1401 HU;
11. Uncontrolled diabetes mellitus (HbA1c >9%).
12. Renal insufficiency.
13. Subjects with arterial hypertension.
14. Subjects with prostate adenoma.
15. Allergy or hypersensitivity to any of the ingredients of the investigational product.
16. BMI ≥ 30 kg/m2.
17. Women who are pregnant or lactating; women who plan on getting pregnant during the study.
18. Alcohol or drug abuse in the last year.
19. Unstable medical conditions, as determined by the Investigator.
20. Inability to comply with the study protocol.
21. Subjects who cannot understand or not capable of completing the study documents.
22. Inability to give informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of subjects without residual fragments or with fragments ≤ 2mm in diameter. | 90 days + 5 days after endourological treatment.
  Percentage of subjects without stones or with fragments ≤ 2mm in diameter 3 months after fURS for laser lithotripsy of kidney stones, assessed by NCCT.

SECONDARY OUTCOMES:
Percentage, size and location of residual fragments. | 90 days + 5 days after endourological treatment.
  The outcome will be categorized by radiologist via NCCT in 2 categories: ≤ 2mm, or > 2mm.
Number of subjects with complications associated with residual fragments or their elimination | at 30 days and 90 days + 5 days after endourological treatment.
  Febrility, renal colic, protracted hematuria, hydronephrosis grade I, II, III, IV.
Percentage of subjects receiving analgesics | Up to 90 days after endourological treatment.
  Administration of antipyretics as reported on the patient diary - YES/NO
Duration of analgesics administration | Up to 90 days after endourological treatment.
  Administration of antipyretics as reported on the patient diary - YES/NO
Severity of pain | Up to 90 days after endourological treatment.
  Clinical assessment of pain is based on visual analogue scale (VAS) from 0 to 10

CONTACTS AND LOCATIONS:
Overall Officials: Marin Georgiev, Prof, PhD, Principal Investigator — UMHAT "Alexandrovska", Head of Department of Urology, Sofia Medical University; Iliya Saltirov, Prof, MD, PhD, DSc, Principal Investigator — Military Medical Academy, Head of Department of Urology and Nephrology; Boyan Atanasov, Prof, PhD, Principal Investigator — UMHAT "Saint Marina", Head of Department of Urology, Medical University of Pleven; Madjid Kadim, Prof, PhD, Principal Investigator — UMHAT "St. George", Head of Department of Urology; Stanislav Valkanov, PhD, Principal Investigator — UMHAT "Kaspela", Department of Urology; Deyan Anakievski, Prof, PhD, Principal Investigator — MHAT "Heart and Brain", Head of Department of Urology; Kaloqn Davidov, Prof, PhD, Principal Investigator — UMHAT "Sofiamed", Head of Department of Urology; Boris Mladenov, PhD, Principal Investigator — UMBALSM "N. I. Pirogov"; Nikolay Kolev, Prof, PhD, Principal Investigator — UMHAT "Dr. Georgi Stranski", Head of Department of Urology; Tosho Ganev, PhD, Principal Investigator — MHAT "St. Anna - Varna",Head of Department of Urology
Locations (9):
- Bulgaria (9):
  - MHAT "Heart and Brain", Burgas
  - UMHAT "Dr. Georgi Stranski", Pleven
  - University Hospital for Active Treatment "Saint Marina", Pleven
  - UMHAT "St. George", Plovdiv
  - UMHAT Kaspela, Plovdiv
  - UMHAT "Alexandrovska", Sofia
  - Military Medical Academy, Sofia
  - UMBALSM "N. I. Pirogov", Sofia
  - UMHAT "Sofiamed", Sofia